CLINICAL TRIAL: NCT01066065
Title: Metabolic Profile and Cardiovascular Biomarker Pattern Compared in naíve Patients Initiating HAART With TDF-FTC and Raltegravir 400mg BID Vs Darunavir 800 mg Plus Ritonavir 100 mg QD; a One Year Follow-up Observational Study
Brief Title: Metabolic Safety of Raltegravir Versus Darunavir in HIV Naive Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Carlos III, Madrid (Other)
Responsible Party: Hospital Carlos III, Vicente Soriano
Other Study IDs: HCIII0110
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-02

CONDITIONS: Cardiovascular Disease; HIV Infections
Keywords: cardiovascular disease; HIV; metabolic disorder; HIV naive patients initiating HAART with Raltegravir or boosted Darunavir
MeSH Terms: conditions — Cardiovascular Diseases; HIV Infections; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Raltegravir Cohort: Patients taking RAL 400 mg BID with Truvada
- Darunavir Cohort: Patients taking Darunavir 800 mg QD plus Norvir 100 mg QD with truvada

SUMMARY:
The advent of new antiretroviral drugs improved the management of HIV naive patients in terms of efficacy. However, the long term metabolic profile of this drugs has not yet been compared and associations between new antiretrovirals and cardiovascular events remains controversial.

Moreover, the better tolerability and easy dosage of this new drugs might hypothetically influence adherence and QOL of HIV patients.

ELIGIBILITY:
Inclusion Criteria:

* VIH-1

Exclusion Criteria:

* pregnancy
* previous Antiretroviral exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive naïve patients regularly attended at a referral outclinic. 1:1 Randomization in two arms by a local electronic process.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
lipid profile defined as a clinically significant increment (delta) in Total cholesterol LDL, HDL y non-LDL cholesterol. | baseline and week 12, 24, 36 and 48
Insulin resistance defined by HOMA index. | baseline and week 12, 24, 36 and 48
Cardiovascular biomarkers: ICAM, VICAM, IL-6, PCR hs... | baseline and week 12, 24, 36 and 48

SECONDARY OUTCOMES:
Antiretroviral adherence and quality of life items. | baseline and week 12,24,36,48
Efficacy defined as viral suppression and CD4 count recovery | baseline and week 12,24,36,48

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Carlos III, Madrid, Spain